CLINICAL TRIAL: NCT01587859
Title: Frequency of True Short Esophagus in Type II-IV Hiatus Hernia
Brief Title: Short Esophagus in Type II-IV Hiatus Hernia
Acronym: SEHH
Status: Completed | Type: Observational
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Sandro Mattioli, Associate Professor, University of Bologna
Other Study IDs: UniboDipTrap
Record Dates: First submitted 2012-04-26; First posted 2012-04-30 (Estimated); Last update posted 2012-04-30 (Estimated); Status verified 2012-04

CONDITIONS: Paraesophageal Hernia
Keywords: esophagus; gastro-esophageal reflux disease; type II-IV hiatal hernia; esophageal surgery; minimally invasive surgery
MeSH Terms: conditions — Hernia, Hiatal; Gastroesophageal Reflux | interventions — Laparoscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cohort: Patients submitted to laparoscopic surgery for Type II-IV hiatus hernia
  Interventions: Procedure: laparoscopic surgery

INTERVENTIONS:
Procedure: laparoscopic surgery — Nissen fundoplication; Collis Gastroplasty.

SUMMARY:
Background:

The existence, diagnosis and treatment of short esophagus is one of the controversies of the past which has recently re-emerged. The missed diagnosis of short esophagus and the consequent inadequacy of treatment is one of the major causes of failure of antireflux surgery.

The daily clinical practice of surgeons dedicated to therapy of esophageal diseases could take advantage of the definition of frequency, preoperative predictors, intraoperative management and post operative outcomes of cases of foreshortened esophagus, in order to offer the patient affected by GERD the elements necessary for a conscious choice of therapy and to plan the best performance of the surgical procedure.

Aims of the Study To define the percentage of cases among the total of antireflux procedures performed for type II-IV hiatus hernia, in which, after standard isolation of the ge junction and dissection of the mediastinal esophagus at least two centimetres of esophagus can not be replaced without any applied tension below the apex of the diaphragmatic hiatus.

DETAILED DESCRIPTION:
The existence, diagnosis and treatment of short esophagus is one of the controversies of the past within esophageal surgery which has recently re-emerged. This entity was described in detail by radiologists in the 60's. Many surgeons confirmed its existence in the operating room, describing the clinical, anatomical and surgical patterns along with the modalities of surgical treatment of shortened esophagus following progressive fibrosis and retraction of the esophageal wall consequent to severe long standing gastro-esophageal reflux disease (GERD). Contrarily other surgeons denied its existence claiming that the gastro-esophageal (GEJ) junction can be reduced into the abdomen without tension in virtually all patients and that the esophagus is, in fact, not shortened. In the case series of open antireflux surgery, the percentage of dedicated procedures aimed to treat the condition of non-reducibility of the GEJ below the diaphragm is highly variable.

In the present era of minimally invasive antireflux surgery, short esophagus again seems to originate controversy and open debate. Many thousands of laparoscopic standard antireflux operations have been performed in the world and numerous articles report satisfactory short and medium-term functional results in over 90% of cases, although in these experiences the need for a tailored approach has not emerged. However, in the last years, many reports on the diagnosis and laparoscopic management of shortened esophagus in GERD surgery have been published.

The perception of "excessive tension" of the fundoplication at the operating table is highly subjective.

During the process of progressive shortening of the esophagus, the portion of the fundus attracted above the diaphragm may take the appearance of a funnel hardly distinguishable from a thickened oesophagus. Therefore the gastric fundus may be erroneously wrapped around the herniated stomach.

Through laparoscopic surgery, by cranially distending the diaphragmatic hiatus the pneumoperitoneum may by artefact increase the length of the intra-abdominal esophagus, and the impossibility to manually palpate and feel the tension applied to the esophagus to bring the GEJ below the diaphragm may make it difficult to recognize a condition of shortened esophagus, more so if the experience of the surgeon is not adequate. The different methods adopted by surgeons in assessing the length and the elasticity of the esophagus and the position of the esophago-gastric junction with respect to the hiatus is the cause of the disagreement. The missed diagnosis of short esophagus and the consequent inadequacy of treatment is one of the major causes of failure of antireflux surgery.

As the number of antireflux operations, mainly laparoscopic, performed per year has remarkably increased, the issue of the so-called short esophagus is today one of the major points in the management of antireflux surgery, which deserves reappraisal and definitive clarification.

The daily clinical practice of surgeons dedicated to therapy of esophageal diseases could take advantage of the definition of frequency, preoperative predictors, intraoperative management and post operative outcomes of cases of foreshortened esophagus in order to offer the patient affected by GERD, the elements necessary for a conscious choice of therapy and to plan the best performance of the surgical procedure.

Aim of this study is: to define the percentage of cases among the total of antireflux procedures performed for type II-IV hiatus hernia, in which, after standard isolation of the GEJ and eventual dissection of the mediastinal esophagus at least two centimetres of esophagus can not be replaced without any applied tension below the apex of the diaphragmatic hiatus; and to record the intra-operative, postoperative outcome of procedures adopted for the surgical treatment of type II-IV hiatus hernia.

ELIGIBILITY:
Inclusion Criteria:

* patients aged > 18 years, undergoing surgery for the treatment of type II-IV hiatus hernia ± GERD, in which a laparoscopic approach is preoperatively indicated.

Exclusion Criteria:

* association of GERD with epiphrenic esophageal diverticulum, collagen diseases, undetermined esophageal motility disorders
* redo antireflux surgery, previous surgery on the thoracic and abdominal esophagus and stomach, on the diaphragm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients consecutively operated upon with minimally invasive surgery for type II-IV hiatus hernia in the period January 1995 - December 2010.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 1995-01; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Global Results | minimum 12 months
  Pre-operatively, patients routinely underwent the symptoms assessment, barium swallow, upper gastro-intestinal endoscopy and esophageal manometry.
  The type and severity of symptoms and the grade of reflux esophagitis were scored using a questionnaire with semi-quantitative scales (form 0 = absence of symptoms or esophagitis, to 3 = severe symptoms and esophagitis.For the surgical results an evaluation scale , from "excellent" to "poor", was used.

CONTACTS AND LOCATIONS:
Overall Officials: Secretary, Principal Investigator — Departement of General Surgery and Organ Transplantation
Locations (2):
- Italy (2):
  - Department of Surgery and Organ Transplantation, Bologna, BO
  - Sandro Mattioli, Bologna, BO

REFERENCES:
- [Derived] Lugaresi M, Mattioli S, Aramini B, D'Ovidio F, Di Simone MP, Perrone O. The frequency of true short oesophagus in type II-IV hiatal hernia. Eur J Cardiothorac Surg. 2013 Feb;43(2):e30-6. doi: 10.1093/ejcts/ezs602. Epub 2012 Nov 27. PMID 23186837